CLINICAL TRIAL: NCT03599700
Title: Risk Factors and Predictors of Thrombosis in Patients With Philadelphia Negative Myeloprolferative Neoplasms
Brief Title: Risk Factors and Predictors of Thrombosis in Myeloprolferative Neoplasms
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maha Mohammed Abdel-Aziz, principal investigator, Assiut University
Other Study IDs: MPN; HABIBA (Other: clinical hematology unit)
Record Dates: First submitted 2018-06-28; First posted 2018-07-26 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Thrombosis
Keywords: thrombosis; myeloproliferative neoplasms
MeSH Terms: conditions — Thrombosis; Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- myeloproliferative neoplasms: * history taking
  * physical examination
  * laboratory investigations: Complete blood counts Bone marrow examination JAK2 V617F mutation. High-sensitivity C-reactive protein ESR Uric acid level LDH GGT BCR- ABL fusion gene IL-8 , TNF-Alpha Serum ferritin Serum albumin, transferrin, alpha feto protein Complement system: C3, C4.
  Interventions: Diagnostic Test: myeloproliferative neoplasms

INTERVENTIONS:
Diagnostic Test: myeloproliferative neoplasms — BLOOD SAMPLING

SUMMARY:
To assess the clinical risk factors and predictable biomarkers of thrombotic complications in cases of philadelphia negative myeloproliferative disorders.

DETAILED DESCRIPTION:
Classic BCR-ABL negative chronic myeloproliferative neoplasms (MPN) are stem cell disorders characterized by abnormal myeloid proliferation and increased blood cell counts and comprise polycythemia vera (PV), essential thrombocythemia (ET) and primary myelofibrosis (PMF).

Myeloproliferative neoplasms (MPN) are common malignancies in elderly individuals as the combined annual incidence rates of classical MPNs were reported to be 0.84, 1.03, and 0.47 per 100,000 respectively for PV, ET, and PMF but with a wide variation in prevalence rates reported in different studies. The 5-year relative survival rates are 84.8, 89.9, and 39% for PV, ET and PMF patients, respectively.

Thromboembolic complications represent a major cause of morbidity and mortality in MPN, particularly in PV and ET. The mechanisms underlying increased thrombotic risk in chronic myeloproliferative neoplasms (MPN) are incompletely understood.

Several pathophysiological mechanisms help explain the increased likelihood of thrombosis in these patients. Factors, such as leukocyte and platelet activation leading to the formation of leukocyte-platelet aggregates, activation of the coagulation cascade by microparticles, high levels of inflammatory cytokines, and endothelial dysfunction have a crucial role in thrombosis in MPN patients.

Accurate prediction of the thrombotic risk still represents a challenge and adequate predictive biomarkers are not available. The mechanisms underlying thrombosis involve a complex interplay among blood cells, the endothelium and the coagulation system. Both increased blood counts and cellular activation, which is due to hyperactivation of intracellular signaling pathways and enhanced interaction between blood cells, are implicated in the thrombotic predisposition.

The JAK2V617F mutation is a diagnostic marker for MPN and it also plays an important role in patient treatment since inhibition of JAK2-associated proliferative pathways has the potential to inhibit cell proliferation in MPNs. This mutation is present in ~95% of PV patients and 50% of ET or PMF patients. Thrombosis and hemostasis are major complications that affect the life expectancy of patients with MPN.

Current guidelines recommend testing for JAK2 mutations in any patient suspected to have an MPN. JAK2 mutation leads to distinct changes in hematopoietic cells that increase the likelihood of thrombus formation.

The risk of thrombosis, in both PV and ET, exceeds 20% and a substantial proportion of patients experience vasomotor disturbances (e.g. headaches, lightheadedness, acral paresthesias, erythromelalgia, atypical chest pain, ocular disturbances, tinnitus) and in case of PV, pruritus.

Mean platelet volume (MPV) is largely considered as a useful indirect marker of platelet activation. Larger platelets are metabolically and enzymatically more active, and have a greater prothrombotic potential. Elevated MPV is associated with other markers of platelet activity, including increased platelet aggregation, increased thromboxane synthesis and beta-thromboglobulin release, and increased expression of adhesion molecules.

High sensitivity CRP is an inflammatory marker might be useful to reflect a condition of chronic inflammation which is associated with the disease severity .

In addition, Elevated CRP and elevated LDH are risk factors for survival in MPN patients.

Elevated γ-Glutamyl (γ-GT) transferase is an independent risk factor for Splanchnic venous thrombosis (SVT) presence in MPN.

About 30% of vascular events in Ph-negative MPN patients are VTE, which generally present as lower limb deep vein thrombosis or pulmonary artery embolism. However, in Ph-negative MPN, VTE characteristically occurs in uncommon locations such as splanchnic veins, including hepatic veins (presenting Budd-Chiari syndrome), portal and mesenteric veins, or, less frequently, cerebral veins or sinuses. In patients with MPN, the prevalence of CVT is 3-7% of cases.

Myeloproliferative neoplasms are known to be pro-thrombotic diseases (arterial and venous). For both of ET and PV, thromboses occur more frequently in arterial sites (between 64 and 75% for PV, and between 72 and 91% for ET).

JAK2 mutation can affect cardiac arteries and veins in ET and PV, which results in thrombosis, ischemia and other cardiovascular events. JAK/STAT signaling pathway plays an important role in heart diseases. High incidence of atrial arrhythmias among patients with ET or PV. The patients were older, cumulating more cardiovascular risk factors inducing more thrombotic events mainly in arteries, and have a higher incidence of death.

The importance of treatment compliance has now been clearly established in many pathological conditions as poor adherence has a negative impact on clinical evolution and non-adherence to cytoreductive therapy was associated with a significant reduction in the complete haematological remission rate but no significant association between thrombosis or death and non-adherence was found. This may be related to the fact that thrombosis is a more acute event, depending on the immediate hemostatic status at the time of thrombus constitution, whereas the phenotypic evolution of chronic haematological malignancies may be more the result of long term evolution of the clone, reflecting its exposure to therapeutic pressure.

Patients with MPN should also avoid factors that are known to increase risk of VTE, including systemic hormone therapy such as oral contraceptive pills and smoking, and optimize cardiovascular risk factors, including control of blood pressure, diabetes, and cholesterol, in order to minimize thrombotic complications.

ELIGIBILITY:
Inclusion Criteria:

age > 18 years

All patients diagnosed as BCR-ABL negative myeloproliferative neoplasm e.g:

Polycythemia vera Essential thrombocythemia Primary myelofibrosis

Exclusion Criteria:

* BCR- ABL positive MPN e.g CML
* Secondary erythrocytosis.
* Secondary thrombocytosis.
* Secondary bone marrow fibrosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: prospective cohort study
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2019-12-20 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of thromboembolic events in Philadelphia negative myeloproliferative neoplasms | 3 years
  Incidence of thromboembolic events e.g. portal vein thrombosis, deep venous thrombosis or pulmonary embolism at patients newly diagnosed as philadelphia negative myeloproliferative neoplasms during the period of the study

SECONDARY OUTCOMES:
survival of patients with Philadelphia negative myeloproliferative neoplasms | 3 years
  life expectancy and causes of death( e.g. thrombosis, bleeding, infections, leukemic transformation)

CONTACTS AND LOCATIONS:
Overall Officials: howida nafady, Study Director — extracted from this organization's records
Locations (1):
- Clinical Hematology Unit, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barbui T, Finazzi G, Falanga A. Myeloproliferative neoplasms and thrombosis. Blood. 2013 Sep 26;122(13):2176-84. doi: 10.1182/blood-2013-03-460154. Epub 2013 Jul 3. PMID 23823316
- [Background] Marin Oyarzun CP, Carestia A, Lev PR, Glembotsky AC, Castro Rios MA, Moiraghi B, Molinas FC, Marta RF, Schattner M, Heller PG. Neutrophil extracellular trap formation and circulating nucleosomes in patients with chronic myeloproliferative neoplasms. Sci Rep. 2016 Dec 13;6:38738. doi: 10.1038/srep38738. PMID 27958278
- [Background] Ball S, Thein KZ, Maiti A, Nugent K. Thrombosis in Philadelphia negative classical myeloproliferative neoplasms: a narrative review on epidemiology, risk assessment, and pathophysiologic mechanisms. J Thromb Thrombolysis. 2018 May;45(4):516-528. doi: 10.1007/s11239-018-1623-4. PMID 29404876
- [Background] Zhang W, Qi J, Zhao S, Shen W, Dai L, Han W, Huang M, Wang Z, Ruan C, Wu D, Han Y. Clinical significance of circulating microparticles in Ph- myeloproliferative neoplasms. Oncol Lett. 2017 Aug;14(2):2531-2536. doi: 10.3892/ol.2017.6459. Epub 2017 Jun 22. PMID 28789461
- [Background] How J, Zhou A, Oh ST. Splanchnic vein thrombosis in myeloproliferative neoplasms: pathophysiology and molecular mechanisms of disease. Ther Adv Hematol. 2017 Mar;8(3):107-118. doi: 10.1177/2040620716680333. Epub 2016 Dec 8. PMID 28246554
- [Background] Tefferi A. Polycythemia vera and essential thrombocythemia: 2013 update on diagnosis, risk-stratification, and management. Am J Hematol. 2013 Jun;88(6):507-16. doi: 10.1002/ajh.23417. PMID 23695894
- [Background] Kissova J, Bulikova A, Ovesna P, Bourkova L, Penka M. Increased mean platelet volume and immature platelet fraction as potential predictors of thrombotic complications in BCR/ABL-negative myeloproliferative neoplasms. Int J Hematol. 2014 Nov;100(5):429-36. doi: 10.1007/s12185-014-1673-0. Epub 2014 Sep 17. PMID 25227185
- [Background] Lussana F, Carobbio A, Salmoiraghi S, Guglielmelli P, Vannucchi AM, Bottazzi B, Leone R, Mantovani A, Barbui T, Rambaldi A. Driver mutations (JAK2V617F, MPLW515L/K or CALR), pentraxin-3 and C-reactive protein in essential thrombocythemia and polycythemia vera. J Hematol Oncol. 2017 Feb 22;10(1):54. doi: 10.1186/s13045-017-0425-z. PMID 28228104
- [Background] Gortzen J, Hunka LM, Vonnahme M, Praktiknjo M, Kaifie A, Fimmers R, Jansen C, Heine A, Lehmann J, Goethert JR, Gattermann N, Goekkurt E, Platzbecker U, Brossart P, Strassburg CP, Brummendorf TH, Koschmieder S, Wolf D, Trebicka J. gamma-Glutamyl Transferase Is an Independent Biomarker of Splanchnic Thrombosis in Patients With Myeloproliferative Neoplasm. Medicine (Baltimore). 2016 May;95(20):e3355. doi: 10.1097/MD.0000000000003355. PMID 27196445
- [Background] Lamy M, Palazzo P, Agius P, Chomel JC, Ciron J, Berthomet A, Cantagrel P, Prigent J, Ingrand P, Puyade M, Neau JP. Should We Screen for Janus Kinase 2 V617F Mutation in Cerebral Venous Thrombosis? Cerebrovasc Dis. 2017;44(3-4):97-104. doi: 10.1159/000471891. Epub 2017 Jun 14. PMID 28609766
- [Background] Mahe K, Delluc A, Chauveau A, Castellant P, Mottier D, Dalbies F, Berthou C, Guillerm G, Lippert E, Ianotto JC. Incidence and impact of atrial arrhythmias on thrombotic events in MPNs. Ann Hematol. 2018 Jan;97(1):101-107. doi: 10.1007/s00277-017-3164-x. Epub 2017 Nov 21. PMID 29164292
- [Background] Haybar H, Khodadi E, Shahjahani M, Saki N. Cardiovascular Events: A Challenge in JAK2-positive Myeloproliferative Neoplasms. Cardiovasc Hematol Disord Drug Targets. 2017;17(3):161-166. doi: 10.2174/1871529X17666171030122345. PMID 29086702
- [Background] Le Calloch R, Lacut K, Le Gall-Ianotto C, Nowak E, Abiven M, Tempescul A, Dalbies F, Eveillard JR, Ugo V, Giraudier S, Guillerm G, Lippert E, Berthou C, Ianotto JC. Non-adherence to treatment with cytoreductive and/or antithrombotic drugs is frequent and associated with an increased risk of complications in patients with polycythemia vera or essential thrombocythemia (OUEST study). Haematologica. 2018 Apr;103(4):607-613. doi: 10.3324/haematol.2017.180448. Epub 2017 Dec 15. PMID 29246923
- [Background] Martin K. Risk Factors for and Management of MPN-Associated Bleeding and Thrombosis. Curr Hematol Malig Rep. 2017 Oct;12(5):389-396. doi: 10.1007/s11899-017-0400-3. PMID 28948496